CLINICAL TRIAL: NCT06777680
Title: Efficacy of Palmitoylethanolamide and Luteolin on Early Functional Recovery in Acute Stroke Patients Treated with Thrombectomy: a Pilot Randomized Placebo-controlled Prospective Study
Brief Title: Palmitoylethanolamide and Luteolin in Patients with Acute Ischemic Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedali Riuniti Trieste (Other)
Responsible Party: Principal Investigator, Marcello Naccarato, Principal Investigator, Ospedali Riuniti Trieste
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: PEALUT - STROKE
Record Dates: First submitted 2025-01-10; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Acute Ischemic Stroke AIS
Keywords: Stroke; Neuroinflammation; Palmitoylethanolamide; Luteolin
MeSH Terms: conditions — Stroke; Neuroinflammatory Diseases | interventions — Luteolin; Thrombectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Active Comparator): co-ultramicronized Palmitoylethanolamide + Luteolin oral suspension (700 mg + 70 mg in 10 ml) in add-on to mechanical thrombectomy
  Interventions: Dietary Supplement: co-ultramicronized Palmitoylethanolamide + Luteolin (770 mg); Procedure: Thrombectomy
- Control group (Placebo Comparator): Placebo oral suspension in add-on to mechanical thrombectomy
  Interventions: Other: Placebo; Procedure: Thrombectomy

INTERVENTIONS:
Dietary Supplement: co-ultramicronized Palmitoylethanolamide + Luteolin (770 mg) — oral suspension, 10 ml twice a day (every 12 hours) for 7 days
  Other Names: Glialia® oral suspension; PEALUT® oral suspension
  Arms: Treatment group
Other: Placebo — oral suspension,10 ml twice a day (every 12 hours) for 7 days
  Arms: Control group
Procedure: Thrombectomy — Endovascular Thrombectomy in all eligible patients, according to national acute stroke treatment guidelines

SUMMARY:
Acute ischemic stroke is caused by reduced blood supply to the brain associated with neuroinflammation. This mechanism contributes to acute neuronal death and persists even after reopening of the closed vessel, with consequent limitation of clinical and functional improvement.

Experimental and clinical evidence demonstrated the anti-inflammatory and neuroprotective effect of micronized and ultramicronized Palmitoylethanolamide (PEA).

The aim of this study is to evaluate the effect of co-ultramicronized PEA and luteolin (700 mg + 70 mg in 10 ml) on the clinical outcomes of patients with acute ischemic stroke undergoing mechanical thrombectomy.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 60 years
* both genders
* first acute ischemic stroke in the middle cerebral artery area confirmed by angio-CT and CTP, eligible for mechanical thrombectomy according to national guidelines
* NIHSS > 6
* compliant patients
* signed informed consent

Exclusion Criteria:

* hemorrhagic stroke
* previous stroke (TIA, ischemic or hemorrhagic stroke)
* presence of clinically evident neurodegenerative diseases (Alzheimer's disease, Parkinson's disease)
* presence of psychiatric comorbidity (schizophrenia, bipolar disorder, depressive syndrome)
* presence of chronic inflammatory diseases (chronic inflammatory bowel disease, vasculitis etc.)
* current or previous neoplasia
* uncontrolled diabetes mellitus (glycemia on admission >400 mg/dL or <50 mg/dL)
* dysphagia, with inability to feed orally
* inability to provide informed consent
* pre-existing disability (pre-stroke mRS >2)
* allergy or hypersensitivity to the study treatment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the mean neurological disability score assessed by National Institutes of Health Stroke Scale (NIHSS), at 3 and 7 days (end of treatment) after hospitalization, between the two groups | Baseline-hospitalization, 3 and 7 days
  NIHSS score ranges from 0 to 42, with higher scores indicating more severe neurological deficit
Change from baseline in the mean functional disability score assessed by modified Rankin Scale (mRS), at 7 days after hospitalization, between the two groups | Baseline-hospitalization and 7 days
  mRS consists of 6 grades from 0 to 5, with 0 corresponding to no symptoms and 5 corresponding to severe disability

SECONDARY OUTCOMES:
Incidence of death and/or major vascular events (recurrent strokes, myocardial ischemia or peripheral arterial ischemia) from baseline to 7 days after hospitalization, between the two groups | From baseline to 7 days
Change from baseline of inflammatory and brain damage mediators [interleukin- 6 (IL-6), matrix metalloproteinase- 9 (MMP-9) and neurofilament light (NfL)] plasma levels at 3 and 7 days after hospitalization, between the two groups | Baseline-hospitalization, 3 and 7 days
Volume of restored penumbra | Baseline-hospitalization, 3 days
  Volume of initial penumbra on admission CT perfusion scans not evolved to ischemic lesion on follow-up CT scan at 72 hrs since stroke onset

CONTACTS AND LOCATIONS:
Overall Officials: Marcello Naccarato, MD, PhD, Principal Investigator — Azienda Sanitaria Universitaria Giuliano Isontina (ASU GI)
Locations (1):
- Azienda Sanitaria Universitaria Giuliano Isontina, Trieste, Italy, Italy

IPD SHARING:
Plan to Share IPD: No